CLINICAL TRIAL: NCT05273320
Title: Phase I Pre-pilot Open-label Clinical Trial of Nabilone for Severe Behavioural Problems (Aggression) in Adults With Intellectual and Developmental Disabilities
Brief Title: Clinical Trial of Nabilone for Aggression in Adults With Intellectual and Developmental Disabilities
Acronym: N-AND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hsiang-Yuan Lin (Other)
Responsible Party: Sponsor-Investigator, Hsiang-Yuan Lin, Clinician-Scientist, Centre for Addiction and Mental Health
Organization: Centre for Addiction and Mental Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135-2020
Record Dates: First submitted 2022-02-11; First posted 2022-03-10 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Intellectual Disability; Developmental Disability; Aggression; Behavior Problem
Keywords: Intellectual Disability; Developmental Disability; Aggression; Behavior Problem
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Aggression; Mental Disorders | interventions — nabilone; Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): Titration: Nabilone p.o., increased in 0.25 mg increments every 2 days to a maximum of 1 mg b.i.d.
  Open label: Nabilone p.o. at maximum dose tolerated for 28 days Tapering: Nabilone p.o. decreased in 0.25 decrements per day
  Interventions: Drug: Nabilone

INTERVENTIONS:
Drug: Nabilone — Nabilone capsules at a maximum dose of 1 mg twice a day
  Other Names: 02392925 Teva-Nabilone 0.25 mg Capsule; 02384892 Teva-Nabilone 1 mg Capsule

SUMMARY:
Innovative treatments are urgently needed for severe behavioural problems (SBPs) in adults with intellectual and developmental disabilities (IDD). Although a synthetic cannabinoid, nabilone may be a plausible and safe alternative to treat SBP, safety and efficacy of nabilone in people with IDD has never been evaluated. The investigators propose to conduct this first-ever Phase I pre-pilot open-label clinical trial to collect data on the tolerability and safety profile of nabilone in adults with IDD, and explore changes in SBP pre- and post-treatment. The results will inform a next-stage pilot randomized controlled trial, followed by a fully powered trial eventually.

DETAILED DESCRIPTION:
Current medications for severe behavioural problems (SBP) show equivocal effectiveness and are associated with a high risk of side effects. Innovative and safe treatments are urgently needed. While preclinical studies, anecdotal reports, and uncontrolled studies link SBP with an endocannabinoid mechanism and suggest that medical cannabinoids may be an efficacious and safe alternative to current medications for SBP in adults with IDD, rigorous evidence is still in the very early stages. Unlike cannabidiol (CBD), a cannabinoid with elusive mechanisms and dose ranges, nabilone, a marketed synthetic cannabinoid, has a clearer mechanism, favourable safety profile, and more predictable dosing. Data of safety and efficacy regarding nabilone in this population has never been published.

This study is a Phase I pre-pilot open-label trial of nabilone in adults with IDD and SBP. The trial first includes a screening visit (S-V) for eligibility, then a baseline visit (V 0), followed by a dose titration phase, and then a 4-week open label phase at a stable dose. At the end of the open label phase, participants will undergo a termination visit (V 1), after which nabilone will be tapered off over 8 days. And then, 2 weeks later, participants will undergo a last follow-up visit (V-F) to ensure safety.

At S-V, and before the informed consent process, the participant will be assessed for capacity to provide informed consent. If they cannot pass the competence test using the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR), then the written informed consent will be obtained from their substitute decision-maker after seeking participants' assent.

At S-V, participants will also be assessed for eligibility based on the inclusion and exclusion criteria, including SBP defined as a score ≥18 on the Aberrant Behaviour Checklist-Irritability subscale (ABC-I) and a score ≥4 on the Clinical Global Impressions-Severity scale. The SBP should present with a consistent pattern with the frequency of ≥1 time per week for >3 months.

At V 0 the following assessments will be completed:

* Clinical Global Impression - Severity scale (CGI-S) will be rated by the investigator to evaluate the severity of the behavioural problems.
* Measuring baseline vital signs and weight to monitor any AEs of nabilone.
* Assessment of participants' cognitive capacity using the NIH Toolbox® Cognition Battery. Previous evidence suggests that nabilone may cause acute mild decrement in attention and working memory. The investigators will use the NIH Toolbox® Cognition Battery, which has been shown as a good candidate outcome measure to examine broad nonverbal cognitive changes for individuals with IDD (valid and reliable for those with a mental age of ≥5 years; implementable for those with a mental age of ≥3 years), to assess the baseline attention and working memory.
* Assessment of SBP of participants, including behavioural problems using the ABC-I and Modified Overt Aggression Scale (MOAS), as reported by the caregivers. These scales will be the principal measures for detection of changes in SBP.
* Assessment of anxiety using the parent-rated General Anxiety Subscale of the Anxiety, Depression, and Mood Scale (ADAMS). Nabilone and THC at low doses have been shown to alleviate anxiety, thus this measure is used for exploratory aims to detect a signal of behavioural/mood change with nabilone use.
* Assessment of caregiver's stress and crisis using the Stress Subscale of Depression Anxiety Stress Scales (DASS-21) and Brief Family Distress Scale (BFDS). As SBP cause major caregiver burden, the investigators aim to assess whether the caregiver's stress and distress would improve if nabilone also improves participants' SBP.
* Exploratory assessment of autism symptoms using the Social Communication Questionnaire for Adults with Intellectual Disability (SCQ-AID). Prior evidence suggests that autistic symptoms may be associated with the presentation of SBP. The investigators aim to explore whether the baseline autistic symptoms would modulate treatment effects of nabilone.
* Optional assessment of MRI Imaging (dependent on the participant's ability to comply with the following assessments, in the opinion of the carers/parents and investigator).

After V 0, eligible participants will receive open-label nabilone starting with a dosage of 0.25 mg before sleep. During the dose titration phase (which could last up to 15 days), nabilone will be titrated in 0.25 mg increments every two days (with the dosing schedule "twice daily") after consultation with the study team during regular phone calls. The study team will also check whether the participants show any physical or mental changes which are believed to be attributed to AEs (based on the UKU side effect rating scale), and advise the participant and their caregivers on the next step of titration accordingly. Dose adjustments are performed until the participant reaches the maximum permitted dose of 1 mg twice daily or experience intolerable AEs believed to be related to nabilone. If intolerable, the participant will use nabilone at the previous lower dose, entering the open label phase.

Participants will be then on a stable, optimized nabilone dosage for four weeks, and then the trial ends with an on-site termination visit (V1). If there are any changes suspected to be associated with AEs, the UKU side effect rating scale will be assessed during the telephone check-up.

At V 1, the following post-treatment assessments will be completed:

* Assessment of adverse events using the UKU side effect rating scale, examined by the researcher or investigator, to systemically investigate the physical AEs of nabilone.
* Re-measuring of vital signs (including blood pressure to check orthostatic hypotension) and weight to monitor the physical AEs of nabilone.
* Re-assessment of participants' cognitive capacity using the NIH Toolbox® Cognition Battery, to monitor any acute cognitive change (AEs) due to nabilone.
* Re-assessment of caregiver rated ABC-I, MOAS, and General Anxiety Subscale of ADAMS. CGI-S and CGI-I will be rated by the investigator to evaluate the severity and improvement of the behavioural problems after nabilone treatment. These re-assessments are implemented to fulfil the exploratory study aim of assessing behavioural changes pre- and post-treatment of nabilone.
* Re-assessment of caregiver's stress and crisis using the Stress Subscale of DASS-21 and BFDS, to investigate changes in their stress and distress after participants takes nabilone.
* Optional re-assessment of MRI Imaging for those who finish the pre-treatment MRI and are willing to receive the second wave of MRI imaging. This is to investigate the change in brain function and structure pre- and post-treatment of nabilone.

Nabilone will be tapered in 0.25 mg daily decrements to prevent acute withdrawal effects. Phone calls will be held every other day during the dose-tapering phase, to check whether there are any changes which are believed to be attributed to withdrawal effects. A safety follow-up visit (S-F) will be scheduled after 2 weeks of full discontinuation from the study drug.

ELIGIBILITY:
Inclusion Criteria:

Participants of any sex or gender, race or ethnicity meeting all criteria listed below will be included in the study:

1. Aged ≥25 years, as medical cannabis should not be used in any person aged <25 as suggested by Health Canada.
2. Adults with a DSM-5 diagnosis of ID meeting: a. Full scale IQ <70 on a standardized cognitive assessment reported in their prior medical record; b. A deficit in adaptive function in at least one activity of life, as estimated by the Adaptive Behavior Assessment System, rated by the caregiver. For those whose verified records are not available, they are deemed eligible if they are connected with Disability Services Ontario. People with ID and other developmental disabilities, e.g., autism, Down syndrome, genetic conditions such as Angelman syndrome, fragile X syndrome, Prader-Willi Syndrome, etc., will also be enrolled.
3. SBP, including aggressive, disruptive, and/or self-injurious behaviours in any situation (home, day program, clinic, etc.), defined as a score ≥18 on the Aberrant Behaviour Checklist-Irritability subscale (ABC-I), and a score ≥4 on the Clinical Global Impressions-Severity scale. A consistent pattern of frequent SBP should occur for >3 months ≥1 time per week.
4. Sexually active women of child-bearing potential must have a negative urine pregnancy test at the screening visit.
5. Sexually active women of child-bearing must use an effective method of birth control at least from the start of last two normal menses before the screening visit to one month after the end of the study (completion of the safety visit). The accepted methods of contraception include total sexual abstinence, if it is the usual and preferred lifestyle, or consistently and correctly taking the oral hormonal contraceptive.
6. Adults who receive a blood test in recent 12 months, which shows liver function test with the ALT ≤3 times the upper limit of normal and bilirubin ≤2 times the upper limit of normal.
7. At least one month that needs to pass from the participation in another investigational drug trial to a given adults being allowed to participate in this trial.

Exclusion Criteria:

1. History of hypersensitivity to any cannabinoid.
2. The presence of an unstable seizure disorder as defined by having not been seizure-free for at least 3 months or anticonvulsant treatment has not been stable for at least 4 weeks.
3. The presence of any clinically significant or unstable medical conditions, including cardiovascular, liver, kidney, pulmonary disease, presence of known congenital brain malformation, as per investigator assessment based on medical history and chart review.
4. The presence of a lifetime diagnosis of psychotic disorders, bipolar disorder, or substance use disorder, or current diagnosis of major depressive disorder or dementia, based on past psychiatric history noted in the medical chart, as well as Moss-PAS (ID) at S-V.
5. Family history of psychotic disorders.
6. Change in psychotropic medications less than 4 weeks prior to study drug use.
7. At the time of screening, each adult's medication list will be checked for drugs that are known to cause interactions with nabilone. When a given adult is taking any drugs or is taking a given medication exceeding a given dose) in the following list, he/she/they will be excluded.

   1. Currently on benzodiazepines at the dose more than the benzodiazepine equivalent to lorazepam 2 mg daily.
   2. Currently on medical psychostimulant, including methylphenidate (100 mg daily), lisdexamfetamine (70 mg daily), amphetamine/dextroamphetamine (Adderall XR®, 50 mg daily), dextroamphetamine (Dexedrine®, 50 mg daily) at the dose exceeding their respective maximum doses (as shown in the bracket after each agent) to treat ADHD in adults, based on the CADDRA guideline, www.caddra.ca.
   3. Currently on nonbenzodiazepine hypnotics, including zaleplon (10 mg daily), zolpidem (10 mg daily), and zopiclone (7.5 mg daily), at the dose exceeding their respective suggested safety doses (as shown in the bracket after each agent), based on Canadian Recalls and Safety Alerts (https://healthycanadians.gc.ca/recall-alert-rappel-avis/).
   4. Currently on any opioids.
   5. Currently on barbiturates.
   6. Drinking any alcohol one week before the screening visit.
   7. Recreational use of any psychomimetic drugs, including Ketamine, LSD, MDMA, Magic mushrooms, PCP, Salvia, GHB, Bath salts, Methamphetamine; the last use happens within one week before the screening visit.
8. Adults currently taking other cannabinoids, such as CBD or medical cannabis, from another source, unless participants and/or their caregivers are willing to stop this treatment for at least 4 weeks prior to entering the study.
9. Adults who might travel out of the area for a significant time during the study.
10. Adults who recently are participating in another investigational drug trial.
11. Pregnancy.
12. Sexually active women of child-bearing potential intended to give breastfeeding or to get pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Physical Adverse Events Assessed by the UKU Side Effect Rating Scale [Safety and Tolerability] | From the titration phase (Week 1) to the safety visit (Week 9)
  Solicited/Unsolicited Physical Adverse Events

OTHER OUTCOMES:
Change From Baseline in Aggression Assessed by Aberrant Behavioral Checklist-Irritability Subscale (ABC-I) at Week 6 | Baseline; Week 6
  Aberrant Behavioral Checklist-Irritability subscale (ABC-I): The ABC is a 58-item rating scale completed by a caregiver. It consists of 5 subscales. Among them, the Irritability subscale consists of 15 items.
Change From Baseline in Aggression Assessed by Modified Overt Aggression Scale (MOAS) at Week 6 | Baseline; Week 6
  Modified Overt Aggression Scale (MOAS) is a reliable measure used to measure behavioural problems in adults with IDD. It consisted of 4 items and is administered by the researcher's interview with the caregiver.
Change From Baseline in Clinician Global Impressions - Severity (CGI-S) Score at Week 6 | Baseline; Week 6
  CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment relative to the clinician's experience with participants who had the same diagnosis. This is rated as: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; or 7 = extremely ill.
Clinical Global Impressions - Improvement (CGI-I) Score at Week 6 | Baseline; Week 6
  CGI-I is a 7-point scale that requires the clinician to assess how much a participant's illness has improved or worsened relative to a Baseline state at the beginning of the intervention. This is rated as: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Yuan Lin, MD, Principal Investigator — Centre for Addiction and Mental Health, Toronto, Ontario, Canada
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No